CLINICAL TRIAL: NCT04952506
Title: A Randomized, Open-label, Single-dosing, 3-treatment, 6-sequence, 3-period, Crossover-design Pilot Clinical Trial to Compare the Safety and Pharmacokinetics of D113 With CKD-349 in Healthy Adult Volunteers
Brief Title: Clinical Study to Compare the Pharmacokinetics and Safety of D113 With CKD-349 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A111_02PK2111P
Record Dates: First submitted 2021-06-29; First posted 2021-07-07 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- R-T1-T2 (Experimental): 1. Period 1: Reference
  2. Period 2: Test 1
  3. Period 3: Test 2
  Interventions: Drug: CKD-349 F1 Tab.; Drug: CKD-349 F2 Tab.; Drug: D113 Tab.
- T2-R-T1 (Experimental): 1. Period 1: Test 2
  2. Period 2: Reference
  3. Period 3: Test 1
  Interventions: Drug: CKD-349 F1 Tab.; Drug: CKD-349 F2 Tab.; Drug: D113 Tab.
- T1-T2-R (Experimental): 1. Period 1: Test 1
  2. Period 2: Test 2
  3. Period 3: Reference
  Interventions: Drug: CKD-349 F1 Tab.; Drug: CKD-349 F2 Tab.; Drug: D113 Tab.
- T2-T1-R (Experimental): 1. Period 1: Test 2
  2. Period 2: Test 1
  3. Period 3: Reference
  Interventions: Drug: CKD-349 F1 Tab.; Drug: CKD-349 F2 Tab.; Drug: D113 Tab.
- T1-R-T2 (Experimental): 1. Period 1: Test 1
  2. Period 2: Reference
  3. Period 3: Test 2
  Interventions: Drug: CKD-349 F1 Tab.; Drug: CKD-349 F2 Tab.; Drug: D113 Tab.
- R-T2-T1 (Experimental): 1. Period 1: Reference
  2. Period 2: Test 2
  3. Period 3: Test 1
  Interventions: Drug: CKD-349 F1 Tab.; Drug: CKD-349 F2 Tab.; Drug: D113 Tab.

INTERVENTIONS:
Drug: CKD-349 F1 Tab. — 1T Single does
  Other Names: Test 1
Drug: CKD-349 F2 Tab. — 1T Single does
  Other Names: Test 2
Drug: D113 Tab. — 1T Single does
  Other Names: Reference

SUMMARY:
This study is a randomized, open-label, single dosing, 3-treatment, 6-sequence, 3-period, crossover-design study to compare the pharmacokinetics and safety of D113 with CKD-349 in healthy volunteers.

DETAILED DESCRIPTION:
To healthy subjects of twenty-four (24), following treatments are administered dosing in each period and wash-out period is a minimum of 7 days.

Reference drug: Entresto 200mg / Test drug: 1) CKD-349 F1 Tab. 2) CKD-349 F2 Tab.

Pharmacokinetic blood samples are collected up to 48hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults over the age of 19 years at the time of screening
2. Individuals who had 18.5 kg/m2 ≤ Body Mass Index(BMI) < 29.9kg/m2 and total body weight ≥ 55 kg

   * BMI = Weight(kg)/ Height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination
4. Individuals who were deemed to be appropriate as study subjects following laboratory tests (hematology, blood chemistry, urinalysis, viral/bacterial, etc.) and vital signs, ECG etc. performed within 28 days to the scheduled date of first administration of the investigational product
5. In case of female subjects, those who were confirmed to be non-pregnant at screening
6. Individuals who agreed to the use of appropriate medically recognized contraceptive methods themselves or their spouse (or partner) from the first administration of the investigational product to the 7th day of last administration. And in case of male subjects, those who agreed not donation of sperm, in case of female subjects, those who agreed not to be pregnant or breast-feeding from the first administration of the investigational product to the 7th day of last administration
7. Individuals who voluntary decide to participate and agrees in writing to comply with the precautions after hearing and fully understanding the detailed explanation of this clinical trial.

Exclusion Criteria:

1. Individuals with a medical evidence or a history of clinically significant hepatobiliary, renal, neurologic, respiratory, digestive, endocrine, blood-oncology, urinary, cardiovascular, musculoskeletal or psychiatric
2. Individuals with symptoms of acute disease within 28 days prior to the scheduled date of first administration of the investigational product
3. Individuals with a medical history of gastrointestinal disease (e.g., Crohn's disease and ulcer) or gastrectomy (excluding simple appendectomy or herniotomy) that may affect drug absorption
4. Individuals with a medical history or current symptoms that fall under one or more of the following who are judged to be concerned about the use of investigational product

   * Individuals with hypersensitivity to investigational products or the investigational products ingredients
   * Angiotensin-converting enzyme(ACE) inhibitors are being administered or less than 36hr after discontinuation.
   * Individuals with history of vascular edema in angiotensin-converting enzyme(ACE) inhibitors or angiotensin receptor blocker(ARB) administration
   * Individuals with genetic or idiopathic angioedema
   * Individuals with liver cirrhosis or atresia of bile ducts or cholestasis
   * Individuals with primary hyperaldosteronism
5. Following vital signs results at screening

   * Sitting systolic blood pressure > 140 mmHg or < 90 mmHg
   * Sitting diastolic blood pressure > 90 mmHg or <60 mmHg
6. Individuals with the following results at screening test:

   * AST(GOT) or ALT(GPT) > 2x the upper limit of the normal range
   * Creatinine > upper limit of the normal range or eGFR with MDRD <60 ml/min/1.73 m2
   * K > 5.5mEq/l
   * Positive reaction on serum test(PRP Ab, anti HIV(AIDS), HBs Ag, HCV Ab)
7. Individuals with a medical history of significant drug abuse or positive for abuse drug in urine test results at screening
8. Individuals who had taken ethical(ETC) or over the counter(OTC) within the 10 days prior to the first dose of investigational product
9. Individuals who donated whole blood within the 8 weeks, or donated blood components within 4 weeks prior to the first dose of the investigational product or received a blood transfusion with 4 weeks
10. Individuals who had been administered investigational product(s) of other clinical study or bioequivalence study within the 6 months prior to the first dose of this study
11. Individuals taking medication known to significantly induce or inhibit drug metabolizing enzymes within 1 month before the first administration of clinical trial drug
12. Individuals who drunk grapefruit juice or caffeine more than 5 cup per day within 3 months prior to first dose of this study or cannot quit drinking during clinical trials period
13. A history of regular alcohol consumption exceeding 21 units/week within the 3 months(1 unit = 10 g = 12.5 ml of pure alcohol) prior to screening or individuals who cannot quit drinking from 48hr prior to the first dose to end of last blooding (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g)
14. Individuals who exceed the smoking amount of 10 cigarettes per day within 3 months prior to first dose of this study or cannot quit smoking during clinical trials period
15. Individuals who cannot eat standard meal in institution
16. Individuals who were deemed to be inappropriate to participate in the study by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-349, D113 | Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  Area under the CKD-349/D113 concentration in blood-time curve from zero to final
Cmax of CKD-349, D113 | Pre-dose (0 hour), post-dose 0.17, 0.33, 0.5, 0.75, 1, 1.33, 1.67, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 48 hours
  The maximum CKD-349/D113 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hee Hong, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No